CLINICAL TRIAL: NCT06463678
Title: A Phase II, Multi-center, Randomized, Masked, Parallel-Control Study to Evaluate the Clinical Efficacy and Safety of IVIEW-1201 (1.0% PVP-Iodine) Gel Forming Ophthalmic Solution in the Treatment of Fungal Keratitis
Brief Title: Trial to Evaluate the Efficacy And Safety of IVIEW-1201 In the Treatment of Fungal Keratitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IVIEW Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IVIEW-1201-FUN- II
Record Dates: First submitted 2024-06-11; First posted 2024-06-18 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Fungal Keratitis
MeSH Terms: interventions — Natamycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IVIEW-1201 (Experimental)
  Interventions: Drug: IVIEW-1201
- NATACYN® (Active Comparator)
  Interventions: Drug: NATACYN®

INTERVENTIONS:
Drug: IVIEW-1201 — Shake well before use and administer 1 drop into the conjunctival sac every 1 hour on Day 1, 2 and 3 when awake; every 2 hours on Day 4-14 when awake; 6 times a day on Day 15-21 with a dosing interval of at least 2.5 hours; 4 times a day on Day 22-28 with a dosing interval of at least 3 hours. The time course of administration is 28 days. After 14 days of dosing, if a patient reaches the primary and secondary endpoints, the investigational drug can be discontinued at the discretion of the investigator.
  Other Names: Treatment Arm
  Arms: IVIEW-1201
Drug: NATACYN® — Shake well before use and administer 1 drop into the conjunctival sac every 1 hour on Day 1, 2 and 3 when awake; every 2 hours on Day 4-14 when awake; 6 times a day on Day 15-21 with a dosing interval of at least 2.5 hours; 4 times a day on Day 22-28 with a dosing interval of at least 3 hours. The time course of administration is 28 days. After 14 days of dosing, if a patient reaches the primary and secondary endpoints, the investigational drug can be discontinued at the discretion of the investigator.
  Other Names: Active Comparator Arm
  Arms: NATACYN®

SUMMARY:
A Phase II, Multi-center, Randomized, Masked, Parallel-Control Study to Evaluate the Clinical Efficacy and Safety of IVIEW-1201 (1.0% PVP-Iodine) Gel Forming Ophthalmic Solution in the Treatment of Fungal Keratitis.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate in the study and signed the Informed Consent Form after receiving a verbal and written explanation of this clinical trial. In cases where the subject is unable to sign the Informed Consent Form, his/her guardian may sign in accordance with relevant regulations.
2. Aged above 15 (inclusive), male or female.
3. Preliminary diagnosis of fungal keratitis based on medical history and clinical observations: corneal focus score ≥ 1.
4. Fungal infection confirmed by laboratory tests (positive for any of the three: fungal hyphae on scraping examination, fungal hyphae on confocal microscopy, positive fungal culture).
5. Not treated with antifungal drugs within 48 hours.
6. Willing to cooperate in the completion of all procedures and visits required for the trial.

Exclusion Criteria:

1. Patients with systemic or ocular diseases, or functional disorders with comorbidities, or structural abnormalities that, in the judgment of the investigator, could adversely affect the course or results of the trial (e.g., hyperthyroidism, hepatitis, acute and chronic renal insufficiency).
2. Those who have a history of allergy or serious adverse reactions to any component of IVIEW-1201 and NATACYN®; a history of allergy or serious adverse reactions to polyene macrolides and other antifungal drugs; or have a cumulative total of three or more allergies to other drugs, food and environment; or have a predisposition to allergic symptoms such as rash or urticaria.
3. Patients with severe cardiac, pulmonary, hepatic, or renal dysfunction and patients with life-threatening or severe unstable underlying diseases.
4. Those with other combined infectious ocular surface diseases.
5. Those with sclera involvement.
6. Those with combined corneal perforation or imminent perforation.
7. Patients with glaucoma and corneal limbal stem cell abnormalities that cannot be cured at the same time, severe chemical burns of cornea and conjunctiva, corneal foreign bodies and other diseases not suitable for this trial.
8. Those who would need to wear corneal contact lenses during the trial.
9. Those who add other medications to treat fungal infections during the trial (except non-facial local treatment).
10. Those who are using other drugs that may interfere with the efficacy or safety evaluation of IVIEW-1201.
11. Systemic use of antifungal drugs within 14 days prior to screening.
12. Systemic use of steroidal drugs within 14 days prior to screening. Local use of eye steroidal drugs or nonsteroidal anti-inflammatory drugs (NSAIDs) within 3 days before enrollment (nasally or bronchially inhaled steroidal drugs are not allowed at any time during the trial).
13. Participation in other interventional clinical trials within 30 days prior to the trial.
14. Pregnant or lactating women, women with positive blood or urine pregnancy tests and those planning to become pregnant (including male subjects); subjects who did not take effective contraceptive measures within 1 month before enrollment, or subjects (including male subjects) who are unwilling to take effective contraceptive measures within the next 6 months.
15. Other conditions or illnesses judged by the clinical investigator to be unsuitable for enrollment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | Day 29 ± 1 day
  Proportion of subjects with a score of 0/12.
  This is manifested by the resolution of clinical symptoms, healing of corneal ulcers, negative fluorescein staining, corneal recovery to translucency or transparency, and resolution of hypopyon.

SECONDARY OUTCOMES:
Fungal clearance | Day 29 ± 1 day
  Positive if fungal hyphae are visible on smear microscopy or confocal microscopy at baseline and negative if no fungal hyphae are visible on smear microscopy or confocal microscopy at the last visit.
Best-corrected visual acuity | Baseline (Day 1) and Day 29 ± 1 day
  The best-corrected visual acuity and its distribution ratio with 0.3, 0.6 and 1.0 LogMAR as cut-offs of test eyes in the test and control groups at baseline and at the last visit. A stratified analysis is carried out to calculate the change in best-corrected visual acuity.